CLINICAL TRIAL: NCT01918995
Title: A Phase 1, Randomized, Double-blind, Dose Escalation, Parallel Group, Placebo-controlled, Repeat Dose Tolerance Study of Regadenoson in Healthy Subjects
Brief Title: Repeat Dose Tolerance Study of Regadenoson in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3606-CL-1005
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Volunteers
Keywords: CVT3146; Regadenoson
MeSH Terms: interventions — regadenoson

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regadenoson low dose (Experimental): Administered over approximately 10 seconds followed by 2 repeat low doses at 10 minute intervals
  Interventions: Drug: Regadenoson
- Regadenoson medium dose (Experimental): Administered over approximately 10 seconds followed by 2 repeat medium doses at 10 minute intervals
  Interventions: Drug: Regadenoson
- Regadenoson high dose (Experimental): Administered over approximately 10 seconds followed by 1 repeat high dose at 10 minute intervals
  Interventions: Drug: Regadenoson
- Placebo (Placebo Comparator): Administered over approximately 10 seconds followed by 1 or 2 repeat doses at 10 minute intervals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regadenoson — Intravenous (IV)
  Other Names: Lexiscan; CVT3146
  Arms: Regadenoson high dose; Regadenoson low dose; Regadenoson medium dose
Drug: Placebo — Intravenous (IV)
  Arms: Placebo

SUMMARY:
This study is to determine the safety, tolerability, and pharmacokinetics of two or three repeat intravenous (IV) bolus doses of regadenoson administered 10 minutes apart in healthy supine subjects.

DETAILED DESCRIPTION:
All subjects will receive up to 3 doses of study drug on day 1 after fasting from all food and drink (except water) for at least 8 hours. Subjects will remain in the clinic for 2 days.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive.
* QTcF must be 430 msec or less for males and 450 msec or less for females. If the mean QTcF exceeds 430 msec for males or 450 msec for females, 1 additional triplicate measurement may be taken. If this triplicate measurement also gives an abnormal QTcF result, the subject should be excluded.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin (TBil) must not be above the normal range. If the Screening test result for AST, ALT, or TBil is > 1 x ULN, but < 1.5 x ULN the assessment may be repeated once during the screening period and on day -1. If the repeat assessment is above the ULN, the subject is not eligible. If the AST, ALT, or TBil test result at Screening is > 1.5 x ULN, it cannot be repeated, and the subject is not eligible.
* Female subject is of non-childbearing potential or if of childbearing potential must use highly effective birth control from Screening through 28 days after the end of the study. Females must not be breastfeeding or donate ova from Screening through 20 days after the end of the study.
* Male subject must be using highly effective contraception from Screening through 90 days after final study drug administration. Male subject must not donate sperm starting at Screening through 90 days after final study drug administration.

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of either Short or Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes).
* The subject has a positive result for hepatitis B surface antigen, hepatitis C antibodies at Screening or is known to be positive for human immunodeficiency virus.
* The subject has a known or suspected allergy to regadenoson or any of the components of the trial products, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions.
* Subject has a history of smoking, regardless of frequency, tobacco type or method of intake, within 6 months prior to first dose of regadenoson.
* The subject has had treatment with any prescribed or non-prescribed drugs in the 2 weeks prior to Day 1, with the exception of occasional use of acetaminophen up to 2 g/day.
* The subject has participated in any interventional clinical study or has received any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to Screening.
* The subject has participated in a prior study with regadenoson.
* The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening or the subject tests positive at screening or Day -1 for alcohol or drugs of abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety assessed by vital signs | Pre-dose and up to 24 hours post dose

SECONDARY OUTCOMES:
Safety assessed by electrocardiogram (ECG), laboratory evaluations, and adverse events | Up to 72 hours after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel Early Phase Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Townsend R, Desai A, Rammelsberg D, Kowalski D, Simmons N, Kitt TM. Safety and tolerability of intravenous regadenoson in healthy subjects: A randomized, repeat-dose, placebo-controlled study. J Nucl Cardiol. 2017 Feb;24(1):57-65. doi: 10.1007/s12350-015-0327-9. Epub 2015 Nov 25. PMID 26607361